CLINICAL TRIAL: NCT04337593
Title: Combination of Basiliximab and Pegaspargase in the Treatment of Relapsed/Refractory Extranodal NK/T-cell Lymphoma, Nasal Type: a Single Arm, Open Label, Phase 2 Trial
Brief Title: Combination of Basiliximab and Pegaspargase in the Treatment of ENKTCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, LIANG WANG, Professor of Department of Hematology, Beijing Tongren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRhos-ENKTCL-4
Record Dates: First submitted 2020-04-04; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Extranodal NK/T-cell Lymphoma
Keywords: extranodal NK/T-cell lymphoma; basiliximab; pegaspargase; CD25
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Basiliximab; PC61 monoclonal antibody; pegaspargase

STUDY DESIGN:
Intervention Model Description: all patients enrolled will received basiliximab and pegaspargase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): 2500 IU/m2 pegaspargase given on day 1, 20 mg basiliximab given on day 1 and 8, repeated every 3 weeks
  Interventions: Drug: Basiliximab; Drug: Pegaspargase

INTERVENTIONS:
Drug: Basiliximab — 20mg d1,8, repeated every 3 weeks
  Other Names: anti-CD25 antibody
Drug: Pegaspargase — 2500IU/㎡, d1,repeated every 3 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Basiliximab in combination with pegaspargase in the treatment of relapsed/refractory NK/T-cell lymphoma.

DETAILED DESCRIPTION:
The investigators previously found that CD25 was elevated in patients who were resistant to chemotherapy, and CD25 can mediate resistance, which can be reversed by targeting CD25 therapy. Thus, the purpose of this study is to evaluate the efficacy and safety of Basiliximab in combination with pegaspargase in the treatment of relapsed/refractory NK/T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathology confirmed diagnosis of NK/T-cell lymphoma.
* Previously treated with pegaspargase-based regimens.
* PET-CT or MRI scan with at least one measurable lesion.
* ECOG score of 0-3 points.
* The lab tests within 1 week before enrollment meets the following:

  * Blood routine: Hb≥80g/L, PLT≥50×10e9/L.
  * Liver function: ALT, AST, TBIL≤2 times the upper limit of normal.
  * Renal function: Cr is normal.
  * Coagulation: plasma fibrinogen≥1.0g/L.
  * Cardiac function: LVEF≥50%, ECG is normal
* Sign the informed consent form.
* Voluntary compliance with research protocols.

Exclusion Criteria:

* Patients with a history of pancreatitis.
* Active infection requires ICU treatment.
* Concomitant HIV infection or active infection with HBV, HCV.
* Serious complications such as fulminant DIC.
* Significant organ dysfunction:

  * respiratory failure
  * NYHA classification≥2 chronic congestive heart failure
  * decompensation Hepatic or renal insufficiency
  * high blood pressure and diabetes that cannot be controlled
  * cerebral vascular events within the past 6 months.
* Pregnant and lactating women.
* Had a history of autoimmune diseases, and disease was active now. Those who were known to be allergic to drugs in the study regimen.
* Patients with other tumors who require treatments within 6 months.
* Other experimental drugs are being used.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
complete response rate | up to 15 weeks±1 week from start of treatment
  evaluated by PET-CT scan or MRI, according to 2014 Lugano criteria for lymphoma

SECONDARY OUTCOMES:
overall response rate | up to 15 weeks±1 week from start of treatment
  evaluated by PET-CT scan or MRI, according to 2014 Lugano criteria for lymphoma
one year progression free survival rate | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Progression free survival was caculated from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first